CLINICAL TRIAL: NCT06350474
Title: A Master Protocol to Test the Impact of Discontinuing Chronic Therapies in People With Cystic Fibrosis on Highly Effective CFTR Modulator Therapy - Dornase Alfa (Dnase)
Brief Title: Impact of Discontinuing Dornase Alfa in People With CF on Highly Effective CFTR Modulator Therapy-A SIMPLIFY Sub-Study
Acronym: SIMPLIFY-DN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nicole Hamblett (Other)
Collaborators: Cystic Fibrosis Foundation (Other); Dartmouth-Hitchcock Medical Center (Other); University of Washington (Other)
Responsible Party: Sponsor-Investigator, Nicole Hamblett, Professor of Pediatrics, Division of Pulmonary and Sleep Medicine, University of Washington School of Medicine Adjunct Professor, Biostatistics, University of Washington School of Medicine Co-Executive Director, Cystic Fibrosis Therapeutics Development, Seattle Children's Hospital
Organization: Seattle Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SIMPLIFY-IP-19 Dnase
Record Dates: First submitted 2024-04-01; First posted 2024-04-05 (Actual); Results first posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; CF; Withdrawal; ETI; dornase alfa; discontinue
MeSH Terms: conditions — Cystic Fibrosis | interventions — Deoxyribonucleases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dnase - Discontinue (Experimental): Discontinuation of current dornase alfa (dnase) therapy
  Interventions: Other: Discontinuation of dornase alfa (Dnase)
- Dnase - Continue (Active Comparator): Continuation of current dornase alfa (dnase) therapy
  Interventions: Other: Continuation of dornase alfa (Dnase)

INTERVENTIONS:
Other: Discontinuation of dornase alfa (Dnase) — Discontinuation of current dornase alfa (Dnase) therapy during 6-week study period.
  Arms: Dnase - Discontinue
Other: Continuation of dornase alfa (Dnase) — Continuation of current dornase alfa (dnase) therapy during 6-week study period. Therapy is taken at least once daily according to each participant's pre-existing, clinically prescribed regimen (e.g., daily, twice daily)
  Arms: Dnase - Continue

SUMMARY:
Despite the increasingly common use of cystic fibrosis transmembrane conductance regulator (CFTR) modulator therapies in treating cystic fibrosis (CF), it is still largely unknown whether or not other chronic therapies can be safely stopped. This SIMPLIFY sub-study is being done to test whether or not it is safe to stop taking dornase alfa (Dnase) in those people that are also taking elexacaftor/tezacaftor/ivacaftor (ETI).

ETI is a combination CFTR modulator therapy that was approved by the Food and Drug Administration for people with CF who have at least one F508del mutation. The three drugs that make up ETI work together to allow many more chloride ions to move into and out of the cells, improving the balance of salt and water in the lungs. These changes result in better clearance of mucus from the lungs and improvements in lung function.

Dornase alfa (Dnase) also improves clearance of mucus from the lungs to support lung function and has been available to people with CF for many years. Dnase is considered to be relatively burdensome and it is not known whether Dnase can improve or maintain lung function above what is already gained through ETI use.

The goal of this SIMPLIFY sub-study is to get information about whether or not it is safe to stop Dnase by testing if there is a change in lung function in participants with cystic fibrosis (CF) who are assigned to stop taking Dnase as compared to those who are assigned to keep taking Dnase while continuing to take ETI.

This is a sub study of master protocol SIMPLIFY-IP-19, NCT04378153.

The sub study investigating the impact of discontinuing and continuing hypertonic saline is registered under NCT06350461.

DETAILED DESCRIPTION:
This SIMPLIFY sub-study (Dornase Alfa (Dnase) Trial) is designed to evaluate the effects of discontinuing Dnase in people with cystic fibrosis (CF) age 12 and older currently taking the highly effective modulator elexacaftor/tezacaftor/ivacaftor (ETI). This is an open label two-arm randomized non-inferiority trial consisting of a 2-week screening period, randomization to continue or discontinue dornase alfa, followed by a 6-week study period. Participants at trial entry will be randomized 1:1 to either continue or discontinue their Dnase therapy.

Clinical outcomes (forced expiratory volume in 1 second [FEV1], antibiotic use, pulmonary exacerbations, and patient reported outcomes), safety (adverse events) and patient reported outcomes to evaluate respiratory symptoms and the participant's perception of how stopping Dnase would impact their daily life will be evaluated in all subjects. Additionally, a subset of participants at selected study sites will participate in Multiple Breath Washout (MBW) to evaluate changes in lung clearance index (LCI).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CF.
* Age ≥ 12 years at the Screening Visit.
* Forced expiratory volume in 1 second (FEV1) ≥ 70 % predicted at the Screening Visit if < 18 years old, and ≥ 60 % predicted at Screening Visit if ≥ 18 years old.
* Clinically stable with no significant changes in health status within the 7 days prior to and including the Screening Visit.
* Current treatment with elexacaftor/tezacaftor/ivacaftor (ETI) for at least the 90 days prior to and including the Screening Visit and willing to continue daily use for the duration of the study.
* Currently taking dornase alfa for at least the 90 days prior to and including the Screening Visit and willing to continue daily use for the 2-week screening period.

Exclusion Criteria:

* Active smoking or vaping.
* Use of an investigational drug within 28 days prior to and including the Screening Visit.
* Changes to chronic therapy (e.g., ibuprofen, azithromycin, inhaled tobramycin, aztreonam lysine) within 28 days prior to and including the Screening Visit. This includes new airway clearance routines.
* Acute use of antibiotics (oral, inhaled or IV) or acute use of systemic corticosteroids for respiratory tract symptoms within 7 days prior to and including the Screening Visit.
* Chronic use of systemic corticosteroids at a dose equivalent to ≥ 10mg per day of prednisone within 28 days prior to and including the Screening Visit.
* Antibiotic treatment for nontuberculous mycobacteria (NTM) within 28 days prior to and including the Screening Visit.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 477 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2022-07-11 (Actual); Study Completion 2022-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Mayer-Hamblett, PhD, Principal Investigator — University of Washington/Seattle Children's; Alex Gifford, MD, FCCP, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (81):
- United States (81):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Tucson Cystic Fibrosis Center, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - CHOC Children's Hospital, Orange, California
  - Stanford University Medical Center, Palo Alto, California
  - Rady Children's Hospital and Health Center at the University of California San Diego, San Diego, California
  - University of California, San Francisco - Adult Center, San Francisco, California
  - University of California, San Francisco - Peds Center, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - National Jewish Health, Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - Nemours Children's Clinic - Jacksonville, Jacksonville, Florida
  - Central Florida Pulmonary Group, Orlando, Florida
  - The Nemours Children's Clinic - Orlando, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Saint Luke's Cystic Fibrosis Center of Idaho, Boise, Idaho
  - Northwestern University, Chicago, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - University of Louisville, Louisville, Kentucky
  - Tulane University, Metairie, Louisiana
  - Maine Medical Partners Pediatric Specialty Care, Portland, Maine
  - John Hopkins Hospital, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan, Michigan Medicine, Ann Arbor, Michigan
  - Wayne State University Harper University Hospital, Detroit, Michigan
  - Corewell Health Helen DeVos, Grand Rapids, Michigan
  - Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - The Minnesota Cystic Fibrosis Center, Minneapolis, Minnesota
  - Children's Mercy Kansas City, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Billings Clinic, Billings, Montana
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Monmouth Medical Center, Eatontown, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Beth Israel Medical Center, New York, New York
  - Lenox Hill Hospital Cystic Fibrosis Center, New York, New York
  - Columbia University Cystic Fibrosis Program, New York, New York
  - University of Rochester Medical Center Strong Memorial, Rochester, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - New York Medical College at Westchester Medical Center, Valhalla, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital/University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cystic Fibrosis Program, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - Oregon Health & Sciences University, Portland, Oregon
  - Hershey Medical Center Pennsylvania State University, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - University of Texas Southwestern / Children's Health, Dallas, Texas
  - University of Texas Southwestern, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - University of Texas Health Center at Tyler, Tyler, Texas
  - Primary Children's Cystic Fibrosis Center, Salt Lake City, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Providence Medical Group, Cystic Fibrosis Center, Spokane, Washington
  - West Virginia University - Morgantown, Morgantown, West Virginia
  - University of Wisconsin, Madison, Wisconsin
  - Children's Wisconsin, Milwaukee, Wisconsin
  - Froedtert & Medical College of Wisconsin, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dnase - Discontinue | Dnase - Continue
Started | 240 | 237
Completed | 238 | 236
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Population: Primary analyses were done on the per-protocol (PP) population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dnase - Discontinue | Dnase - Continue | Total
Number analyzed (Participants) | 199 | 193 | 392
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.1 (9.39) | 23.7 (11.83) | 22.9 (10.7)
Age, Customized [Count of Participants; unit: Participants]
  Age Distribution (years): >=12 to <18 | 89 | 85 | 174
  Age Distribution (years): >=18 to <24 | 45 | 36 | 81
  Age Distribution (years): >=24 to <30 | 25 | 27 | 52
  Age Distribution (years): >=30 | 40 | 45 | 85
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 97 | 195
  Male | 101 | 96 | 197
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 192 | 187 | 379
  Race: Black or African American | 1 | 3 | 4
  Race: Asian | 0 | 1 | 1
  Race: American Indian or Alaskan Native | 1 | 0 | 1
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Race: Other, More than One Race, or Unknown/Not Reported | 5 | 2 | 7
Cystic Fibrosis (CF) Genotype [Count of Participants; unit: Participants]
  F508del Homozygous | 105 | 115 | 220
  F508del Heterozygous | 90 | 73 | 163
  Other or Unknown | 4 | 5 | 9
Forced Expiratory Volume in 1 second (FEV1) [Mean (Standard Deviation); unit: liters] | 3.3 (0.88) | 3.3 (0.86) | 3.3 (0.87)
FEV1 (% Predicted) [Mean (Standard Deviation); unit: percent predicted] — FEV1 % predicted is calculated using the Global Lung Initiative multi-ethnic reference equations for ages 3-95.
  percent predicted | 96.8 (17.40) | 97.0 (16.35) | 96.9 (16.87)
FEV1 (% Predicted) Distribution [Count of Participants; unit: Participants] — Measure Description: FEV1 % predicted is calculated using the Global Lung Initiative multi-ethnic reference equations for ages 3-95.
  Participants
    <60 | 1 | 3 | 4
    >=60 to <70 | 16 | 10 | 26
    >=70 to <90 | 46 | 48 | 94
    >=90 to <100 | 42 | 42 | 84
    >=100 | 94 | 90 | 184
Current Dornase Alfa Use [Count of Participants; unit: Participants] — Use as reported at screening prior to randomization.
  Participants | 199 | 193 | 392
Current Airway Clearance Use [Count of Participants; unit: Participants] — Includes airway clearance by route chest PT/vest.
  Participants | 187 | 185 | 372

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in FEV1 % Predicted From Week 0 to Week 6
Description: Non-Inferiority statistical testing compared difference between study arms (discontinue - continue) in the absolute change in FEV1 % predicted from Week 0 to Week 6.
Time Frame: Week 0 to Week 6
Population: Per-protocol (PP) population.
Measure: Mean (Standard Deviation); unit: FEV1 % predicted
Arm/Group | Dnase - Discontinue | Dnase - Continue
Number analyzed (Participants) | 199 | 193
FEV1 % predicted | 0.2 (3.69) | -0.2 (4.37)
Statistical Analysis 1: Comparison: Dnase - Discontinue vs Dnase - Continue; The non-inferiority test was a priori designed to be conducted on the per-protocol (PP) population; Test type: Non-Inferiority — The non-inferiority margin is -3; p < 0.0001, ANOVA — One-sided test for non-inferiority; Adjusted for four dichotomous randomization strata; Mean Difference (Final Values) = 0.346, 95% CI 2-sided [-0.5 to 1.1] — Direction of difference is Discontinue - Continue

2. Secondary Outcome: Absolute Change in LCI 2.5 From Baseline to Week 6
Description: Statistical testing compared difference between study arms (discontinue - continue) in the absolute change in LCI 2.5 (Lung Clearance Index) from Baseline (Week 0, if available, or else Week -2) to Week 6. LCI 2.5 is the number of times the volume in the lungs needs to turn over to expel an inert gas. A higher value of LCI 2.5 indicates poorer lung function.
Time Frame: Baseline (Week 0 or Week -2) to Week 6
Population: Participants in the per-protocol (PP) population with an acceptable LCI 2.5 measurement at baseline and at Week 6.
Measure: Mean (Standard Deviation); unit: number of lung volume turnovers
Arm/Group | Dnase - Discontinue | Dnase - Continue
Number analyzed (Participants) | 40 | 42
number of lung volume turnovers | -0.1 (0.63) | 0.0 (0.56)
Statistical Analysis 1: Comparison: Dnase - Discontinue vs Dnase - Continue; Test type: Superiority; p = 0.414, ANOVA; Adjusted for four dichotomous randomization strata; Mean Difference (Final Values) = -0.11, 95% CI 2-sided [-0.4 to 0.2] — Direction of difference is Discontinue - Continue

3. Secondary Outcome: Absolute Change in Respiratory Symptoms, as Measured by the CF Respiratory Symptoms Diary-Chronic Respiratory Infection Symptom Severity Score (CRISS) From Week 0 to Week 6
Description: Statistical testing compared the difference between study arms (discontinue - continue) in the absolute change in respiratory symptoms, as measured by the CF Respiratory Symptoms Diary-Chronic Respiratory Infection Symptom Severity Score (CRISS) from Week 0 to Week 6. The Cystic Fibrosis Respiratory Symptoms Daily Diary (CFRSD) asks a participant to state the extent of their 8 respiratory symptoms: difficulty breathing, feverishness, tiredness, chills or sweats, coughing, coughing up mucus, tightness in the chest and wheezing. Each respiratory symptom is assigned a score from 0-4 based on the response, with zero corresponding to the absence of the symptom and four corresponding to symptom being present 'a great deal' or 'extremely'. A summed score (range from 0-24) is calculated for each participant and converted to a final score with a range of 0 to 100 where the lowest scores indicate improvement of symptoms. Calculation of a score requires responses for at least 7 out of 8 symptoms
Time Frame: Week 0 to Week 6
Population: Participants in the per-protocol (PP) population with a CRISS score at Week 0 and at Week 6.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dnase - Discontinue | Dnase - Continue
Number analyzed (Participants) | 199 | 193
score on a scale | -0.1 (9.49) | -1.1 (10.21)
Statistical Analysis 1: Comparison: Dnase - Discontinue vs Dnase - Continue; Test type: Superiority; p = 0.241, ANOVA; Adjusted for four dichotomous randomization strata; Mean Difference (Final Values) = 0.95, 95% CI 2-sided [-1.0 to 2.9] — Direction of difference is Discontinue - Continue

4. Secondary Outcome: Absolute Change in Respiratory Symptoms, as Measured by CFQ-R Respiratory Domain From Week 0 to Week 6
Description: Statistical testing compared the difference between study arms (discontinue - continue) in the absolute change in respiratory symptoms, as measured by the Cystic Fibrosis Questionnaire-Revised Respiratory Domain Score from Week 0 to Week 6. The Cystic Fibrosis Questionnaire - Revised asks participants 6 questions related to respiratory symptoms which are each assigned a score 1-4. The Respiratory Domain Scaled Score is calculated as follows: 100*[{sum of responses}/{number of responses}-1]/3 only if number of responses ≥ 3; otherwise the score is set to missing. The scaled score ranges from 0 to 100 where higher scores indicate improvement of symptoms.
Time Frame: Week 0 to Week 6
Population: Participants in the per-protocol (PP) population with a score at Week 0 and at Week 6.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dnase - Discontinue | Dnase - Continue
Number analyzed (Participants) | 198 | 191
score on a scale | -0.9 (6.23) | 0.0 (8.85)
Statistical Analysis 1: Comparison: Dnase - Discontinue vs Dnase - Continue; Test type: Superiority; p = 0.233, ANOVA; Adjusted for four dichotomous randomization strata; Mean Difference (Final Values) = -0.92, 95% CI 2-sided [-2.5 to 0.6] — Direction of difference is Discontinue - Continue

5. Secondary Outcome: Absolute Change in FEV1 % Predicted From Week -2 to Week 0
Description: Statistical testing compared the difference between study arms (discontinue - continue) in the absolute change in FEV1 % predicted from Week -2 to Week 0.
Time Frame: Week -2 to Week 0
Population: Per-protocol (PP) population.
Measure: Mean (Standard Deviation); unit: FEV1 % predicted
Arm/Group | Dnase - Discontinue | Dnase - Continue
Number analyzed (Participants) | 199 | 193
FEV1 % predicted | 0.2 (3.11) | 0.0 (3.79)
Statistical Analysis 1: Comparison: Dnase - Discontinue vs Dnase - Continue; Test type: Superiority; p = 0.42, t-test, 2 sided; Mean Difference (Final Values) = 0.28, 95% CI 2-sided [-0.4 to 0.97] — Direction of difference is Discontinue - Continue

6. Secondary Outcome: Absolute Change in FEV1 % Predicted From Week 0 to Week 2
Description: Statistical testing compared the difference between study arms (discontinue - continue) in the absolute change in FEV1 % predicted from Week 0 to Week 2.
Time Frame: Week 0 to Week 2
Population: Participants in the per-protocol (PP) population with FEV1 measurements at Week 0 and at Week 2.
Measure: Mean (Standard Deviation); unit: FEV1 % predicted
Arm/Group | Dnase - Discontinue | Dnase - Continue
Number analyzed (Participants) | 196 | 189
FEV1 % predicted | -0.1 (3.67) | 0.1 (3.96)
Statistical Analysis 1: Comparison: Dnase - Discontinue vs Dnase - Continue; Test type: Superiority; p = 0.69, t-test, 2 sided; Mean Difference (Final Values) = -0.15, 95% CI 2-sided [-0.92 to 0.61] — Direction of difference is Discontinue - Continue

7. Secondary Outcome: Number and Percent of Participants Initiating Acute Antibiotics From Week 0 to Week 6
Description: Difference between study arms (discontinue - continue) in the percent of subjects initiating acute oral, inhaled or intravenous antibiotics from Week 0 to Week 6. Includes antibiotics initiated for respiratory indications; excludes those taken as part of a chronic cycled regimen or for a UTI, skin infection, etc.
Time Frame: Week 0 to Week 6
Population: Intent-to-treat (ITT) population of all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Dnase - Discontinue | Dnase - Continue
Number analyzed (Participants) | 240 | 237
Participants | 14 | 8
Statistical Analysis 1: Comparison: Dnase - Discontinue vs Dnase - Continue; Test type: Superiority; p = 0.275, Fisher Exact; Difference in % Participants = 2.5, 95% CI 2-sided [-1.5 to 6.5] — Confidence interval calculated using the Newcombe-Wilson method without continuity correction. Direction of difference is Discontinue - Continue

8. Secondary Outcome: Number and Percent of Participants Hospitalized From Week 0 to Week 6
Description: Statistical testing compared the difference between study arms (discontinue - continue) in the percent of subjects hospitalized from Week 0 to Week 6.
Time Frame: Week 0 to Week 6
Population: Intent-to-treat (ITT) population of all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Dnase - Discontinue | Dnase - Continue
Number analyzed (Participants) | 240 | 237
Participants | 0 | 0

9. Secondary Outcome: Number and Percent of Participants Experiencing Pulmonary Exacerbations From Week 0 to Week 6
Description: Statistical testing compared the difference between study arms (discontinue - continue) in the percent of subjects experiencing a pulmonary exacerbation from Week 0 to Week 6. Pulmonary exacerbations defined using Fuchs criteria.
Time Frame: Week 0 to Week 6
Population: Intent-to-treat (ITT) population of all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Dnase - Discontinue | Dnase - Continue
Number analyzed (Participants) | 240 | 237
Participants | 4 | 2
Statistical Analysis 1: Comparison: Dnase - Discontinue vs Dnase - Continue; Test type: Superiority; p = 0.686, Fisher Exact; Difference in % Participants = 0.8, 95% CI 2-sided [-1.6 to 3.4] — [estimate comment as in outcome 7, analysis 1]

10. Secondary Outcome: Number and Percent of Participants Experiencing Adverse Events (AEs) From Week 0 to Week 6
Description: Statistical testing compared the difference between study arms (discontinue - continue) in the percent of participants with at least one AE from Week 0 to Week 6. Includes serious and non-serious AEs.
Time Frame: Week 0 to Week 6
Measure: Count of Participants; unit: Participants
Arm/Group | Dnase - Discontinue | Dnase - Continue
Number analyzed (Participants) | 240 | 237
Participants | 89 | 55
Statistical Analysis 1: Comparison: Dnase - Discontinue vs Dnase - Continue; Null hypothesis: proportion of participants with at least one AE is the same in Discontinue and Continue arms; Test type: Superiority; p = 0.0010, Fisher Exact; Difference in % Participants = 13.9, 95% CI 2-sided [5.6 to 21.8] — [estimate comment as in outcome 7, analysis 1]

11. Secondary Outcome: Rate of Adverse Events (AEs) From Week 0 to Week 6 Therapy Arms
Description: Statistical testing compared the compared the rate of AE occurrence (number of events divided by total follow-up weeks in each arm) between study arms from Week 0 to Week 6. Includes serious and non-serious AEs.
Time Frame: Week 0 to Week 6
Population: Intent-to-treat (ITT) population of all randomized participants.
Measure: Number; unit: events per week
Arm/Group | Dnase - Discontinue | Dnase - Continue
Number analyzed (Participants) | 240 | 237
events per week | 0.116 | 0.060
Statistical Analysis 1: Comparison: Dnase - Discontinue vs Dnase - Continue; Rate ratio, confidence interval, and p-value calculated using Poisson Regression with an offset for the log of follow-up time in weeks. The total number of follow-up weeks in the DA-discontinue and DA-continue arms are 1486.3 and 1471.4 weeks, respectively. Ratio is Discontinue / Continue; Test type: Superiority; p < 0.0001, Poisson Regression; Rate Ratio = 1.95, 95% CI 2-sided [1.51 to 2.53]

12. Secondary Outcome: Number and Percent of Participants With Temporary or Permanent Changes From Assigned Therapy Regimen Due to Adverse Event From Week 0 to Week 6
Description: Statistical testing compared the difference between study arms (discontinue - continue) in the percent of subjects temporarily or permanently changing their assigned therapy regimen due to an adverse event Week 0 to Week 6
Time Frame: Week 0 to Week 6
Population: Intent-to-treat (ITT) population of all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Dnase - Discontinue | Dnase - Continue
Number analyzed (Participants) | 240 | 237
Participants | 7 | 2
Statistical Analysis 1: Comparison: Dnase - Discontinue vs Dnase - Continue; Null hypothesis: proportion of participants changing assigned regimen is the same in Discontinue and Continue arms; Test type: Superiority; p = 0.1758, Fisher Exact; Difference in % Participants = 2.03, 95% CI 2-sided [-0.6 to 5.0] — [estimate comment as in outcome 7, analysis 1]

ADVERSE EVENTS:
Time Frame: From randomization (Week 0) up to last study visit (Week 6), i.e., 6 weeks.
Arm/Group | Dnase - Discontinue | Dnase - Continue
All-Cause Mortality (participants affected / at risk) | 0/240 | 0/237
Serious Adverse Events (participants affected / at risk) | 0/240 | 0/237
Other Adverse Events (participants affected / at risk) | 25/240 | 14/237
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dnase - Discontinue (N=240) | Dnase - Continue (N=237)
Cough (Respiratory, thoracic and mediastinal disorders) | 16 (16) | 10 (10)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-02-14): https://cdn.clinicaltrials.gov/large-docs/74/NCT06350474/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-06): https://cdn.clinicaltrials.gov/large-docs/74/NCT06350474/SAP_001.pdf